CLINICAL TRIAL: NCT01418937
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK-580299) in Healthy Female Control Subjects From the GSK HPV-023 Study
Brief Title: Safety Evaluation of a Human Papillomavirus (HPV) Vaccine in Healthy Female Control Subjects From the GSK HPV 023 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 114379
Record Dates: First submitted 2011-08-12; First posted 2011-08-17 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine; serious adverse events (SAEs); medically significant conditions; cervical neoplasia
MeSH Terms: conditions — Papillomavirus Infections

ARMS (1):
- HPV Group (Experimental)
  Interventions: Biological: CervarixTM (GSK580299)

INTERVENTIONS:
Biological: CervarixTM (GSK580299) — Three intramuscular injections

SUMMARY:
This phase IIIb study is designed to assess the safety of GlaxoSmithKline Biological's HPV vaccine GSK580299 in female subjects who took part in the HPV-023 (NCT00518336) study and received a placebo in the HPV-001 (NCT00689741) study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A subject previously enrolled in Study HPV-023 (NCT00518336), who received placebo in Study HPV-001 (NCT00689741), and who is 26 years of age or older.
* Written informed consent must be obtained from the subject prior to enrollment.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or breastfeeding: enrollment should be deferred to at least three months after delivery and after breastfeeding is ceased.
* A woman planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase of the study, and up to two months after the last vaccine dose.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen in the protocol.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of each dose of the vaccine, with the exception of administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine. Enrollment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous administration of vaccine components.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Cancer or autoimmune disease under treatment.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrollment. Enrollment will be deferred until condition is resolved.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, which in the opinion of the investigator precludes administration of the study vaccine.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2012-05-29; Primary Completion 2015-01-09 (Actual); Study Completion 2015-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Brazil (5):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Cervarix Group: Subjects received 3 intramuscular injections of Cervarix™ vaccine according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 164
Completed | 156
Not Completed | 8
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 1
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the study period (from Month 0 up to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 164
Subjects
  Any SAEs | 1
  Grade 3 SAEs | 1
  Related SAEs | 0

2. Primary Outcome: Number of Subjects With Potential Immune-mediated Disease (pIMDs)
Time Frame: Throughout the study period (from Month 0 up to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 164
Subjects
  Any pIMDs | 0
  Grade 3 pIMDs | 0
  Related pIMDs | 0

3. Primary Outcome: Number of Subjects With Medically Significant Conditions (MSCs)
Description: MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Throughout the study period (from Month 0 up to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 164
Subjects
  Any MSCs | 8
  Grade 3 MSCs | 1
  Vaccine-related MSCs | 0

4. Primary Outcome: Number of Pregnant Subjects Reporting Pregnancy Outcomes
Description: The pregnancy outcomes were based on reports from pregnant subjects in the study population. Pregnancy outcomes are pregnancies resulting in live births.
Time Frame: Throughout the study period (from Month 0 up to Month 12)
Population: The analysis was performed on the number of pregnant subjects participating in the study.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 5
Subjects | 5

ADVERSE EVENTS:
Time Frame: SAEs were collected throughout the entire study period (from Day 0 to Month 12)
Description: Non-serious solicited and unsolicited adverse events were not collected in this study.
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 1/164
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=164)
Depression suicidal (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.